CLINICAL TRIAL: NCT05450666
Title: Effectiveness of Mobility Exercises in Resistance-Trained Males With Shoulder Immobility in Different Age Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Effectiveness of Mobility Exercises in Resistance-Trained Males with Shoulder Immobility in Different Age Groups, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hazal genç 3
Record Dates: First submitted 2022-07-04; First posted 2022-07-11 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Mobility Limitation; Exercises
Keywords: exercise; body builders
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Intervention Model Description: Evaluation was made before the exercise application, after the eight-week application.
Who Masked: Investigator
Masking Description: Treatment and evaluation in the study were performed by different physiotherapists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YOUNG GROUP (Experimental): The same exercise program will be applied to both groups. Participants will be included in the exercise program for eight weeks. Athletes between the ages of 18 and 30 will be included in this group.
  Interventions: Other: mobility exercises
- ADULT GROUP (Experimental): The same exercise program will be applied to both groups. Participants will be included in the exercise program for eight weeks. Athletes between the ages of 30 and 60 will be included in this group.
  Interventions: Other: mobility exercises

INTERVENTIONS:
Other: mobility exercises — Before starting the exercise program, a video and exercise program including the importance of shoulder mobilization and stabilization and the knowledge of how to contract the right muscle groups will be shared in order to raise awareness of the athletes. Following the evaluations, in addition to the classical training programs, the athletes will perform the Wall Angels and Anterior Shoulder Stretch, Shoulder Circle Rotation, Prone Shoulder Controlled Articular Rotations and Shoulder Side Stretch exercises, Prone I, T, W, Y's 3 days a week for 8 weeks, accompanied by the same physiotherapist.

SUMMARY:
The shoulder is a dynamic and mobile joint between the arm and the trunk. The movement of the joint in three dimensions performs complex movements in almost every activity of daily life.

These movements performed during activities of daily living can cause musculoskeletal problems and shoulder pathologies. For this reason, the shoulder joint should be carefully evaluated, especially in athletes.

DETAILED DESCRIPTION:
The shoulder consists of four functional joints. Glenohumeral joint (GH), acromioclavicular joint (AC), sternoclavicular joint (SC), and scapulothoracic joint (ST). The most mobile of these four joints is the glenohumeral joint, located between the scapula and the glenoid. The GH is a synovial joint that has three-dimensional motion, covers the intra-articular capsule, and wraps the biceps long head tendon to the biceps sulcus. The glenohumeral capsule, glenohumeral ligament, and coracohumeral ligament contain a capsuloligamentous complex structure. This complex structure and the rotator cuff tendons form a static and dynamic restrictive structure around the glenohumeral joint. The rotator cuff space forms a triangular tissue between the edge of the anterior supraspinatus tendon and the superior subscapularis, and the apex is located on the lateral ridge of the biceps sulcus at the edge of the humeral ligament.

After providing mobility, movement and balance will return to stability. Increasing muscle strength for joint stabilization is a physical training goal for the shoulder in athletes.

Bone mechanics, intra-articular pressure, glenohumeral labrum and capuloligamentous structures are static components.

Dynamic components are provided by muscle activity coordinated around the joint and modulated by the neuromuscular system.

The basis of static and dynamic interactions is mainly proprioceptive inputs that occur with mechanoreceptors in the muscles, joint capsule ligaments, tendons and skin, which are integrated into each other.

Joint stabilization is provided by the coactivation force of dynamic shoulder stabilizers.

The balance of such forces must be proportional. For this reason, exercises to provide joint stabilization should aim to provide equal force distribution around the joint.

Among the criteria for evaluating the athletes; proprioception and range of motion.

Body Awareness Questionnaire aims to evaluate body awareness. Posture will be evaluated with New York posture analysis.

As a result of the literature review carried out; As far as is known, there is no adequate, up-to-date and evidence-based study in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Resistance-trained males over the age of 18 with shoulder immobility.

Exclusion Criteria:

* The criteria for exclusion from the study were: having orthopedic or neurological problems, and having undergone upper extremity musculoskeletal surgery.

  * Female resistance-trained,
  * Athletes under the age of 18 will not be included in the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Body Awareness Questionnairei | 8 weeks
  Body awareness basically refers to an individual's awareness of body parts. Body awareness measurement provides the definition of body awareness and evaluation of the effectiveness of the exercise programs to be applied. Body Awareness Questionnaire is a questionnaire consisting of four subgroups (changes in body process, sleep-wake cycle, prediction at the onset of the disease, prediction of body responses) and a total of 18 statements, which are conducted to determine the normal or abnormal sensitivity level of body components. Individuals are asked to score between 1 and 7 for each statement. Grading is done on the total score. A high score indicates that the individual's body sensitivity is good.
The range of motion | 8 weeks
  The range of motion of the shoulder flexion, abduction, internal and external rotator muscles will be measured with a goniometer. Measurements will be made by the dominant side of the athlete in evaluations other than bilateral functional tests. Joint range of motion assessment was measured with a goniometer

SECONDARY OUTCOMES:
New York Posture Scale | 8 weeks
  Posture is the state of being in the most suitable position of every part of the body in relation to the adjacent segment and the whole body.
  Posture analysis is done while standing upright. The postures of the subjects participating in the study were evaluated with the New York Posture Scale. In this evaluation system, posture that can occur in 13 different parts of the body is evaluated. For scoring, a score of five was given if the person's posture was correct, three if it was moderately impaired, and one if it was severely impaired. The total score obtained with the test evaluation is a maximum of 65 and a minimum of 13. The standard evaluation criteria developed for this test were defined as "very good" if the total score is >=45, "good" if 40-44, "moderate" if 30-39, "poor" if 20-29, and "poor" if <=19. detected.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salles JI, Costa F, Cunha-Cruz V, Cagy M, Piedade R, Ribeiro P. Electrophysiological analysis of the perception of passive movement. Neurosci Lett. 2011 Aug 26;501(2):61-6. doi: 10.1016/j.neulet.2011.05.005. Epub 2011 May 7. PMID 21596095
- [Background] Moro T, Tinsley G, Bianco A, Marcolin G, Pacelli QF, Battaglia G, Palma A, Gentil P, Neri M, Paoli A. Effects of eight weeks of time-restricted feeding (16/8) on basal metabolism, maximal strength, body composition, inflammation, and cardiovascular risk factors in resistance-trained males. J Transl Med. 2016 Oct 13;14(1):290. doi: 10.1186/s12967-016-1044-0. PMID 27737674